CLINICAL TRIAL: NCT03658655
Title: Open, One-arm, Single-center Clinical Study to Evaluate the Efficacy and Safety of Stem Cells From Human Exfoliated Teeth in the Treatment of Type 2 Diabetes
Brief Title: Stem Cells From Human Exfoliated Teeth in Treatment of Type 2 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CAR-T (Shanghai) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTLC001
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-10

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem Cells From Human Exfoliated Teeth (Experimental): According to the weight of 0.1IU /kg with Stem Cells From Human Exfoliated Teeth, three injections will be given respectively at the time of enrollment, one week and four weeks after enrollment.
  Interventions: Biological: Stem Cells From Human Exfoliated Teeth

INTERVENTIONS:
Biological: Stem Cells From Human Exfoliated Teeth — Basic treatment:
  The original treatment regimen will be maintained during the study period, insulin dose could be adjusted with the change of blood glucose, while the type and dose of oral hypoglycemic drugs remained unchanged (except when side effects of drugs or insulin preparations were stopped, but patients still had frequent hypoglycemia).
  Stem cell therapy:
  Usage: drip slowly, 50ml normal saline first, then Stem Cells From Human Exfoliated Teeth (during 60 min), then 50ml normal saline.

SUMMARY:
To evaluate the safety and efficacy of Stem Cells From Human Exfoliated Teethtransplantation in patients with type 2 diabetes to provides scientific basis for further clinical studies to verify the safety and efficacy of type 2 diabetes.On the basis of maintaining the original treatment, intravenous drip of Stem Cells From Human Exfoliated Teeth.

DETAILED DESCRIPTION:
Basic treatment:

The original treatment regimen was maintained. During the study period, insulin dose could be adjusted with the change of blood glucose, while the type and dose of oral hypoglycemic drugs remained unchanged (except when side effects of drugs or insulin preparations were stopped or patients still had frequent hypoglycemia).

Stem cell therapy:

Dosage: Stem Cells From Human Exfoliated Teeth were calculated at 0.1IU/kg body weight .

Course of treatment: 3 times, respectively at the time of enrollment, 1 week after enrollment and 4 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the purpose of clinical trial, voluntarily participate in and sign the informed consent;
* Patients with type 2 diabetes WHO were clearly diagnosed according to WHO diagnostic criteria with a course of over 5 years;
* Fasting blood glucose (FPG) was still 7.5-12.0mmol/L and hemoglobin a1c (HbAlc) was still 7.0-10.0% after insulin treatment or combined with oral hypoglycemic drugs; Among them, insulin has been treated for 1 year, and the number of subcutaneous injection is 2 times or more in the last 3 months, and the type and dose of oral hypoglycemic drugs (including metformin only, antinylglycosidase inhibitors or insulin prolactin) have been stable and decreased for 3 months.
* Age 45 to 65 years male and female;
* Body mass index (BMI) between 20 and 30kg/m2;
* Male or Female subjects of childbearing age shall voluntarily take birth control measures from the screening date to the end of the follow-up;Urine pregnancy test was negative during screening of women of reproductive age, and serum pregnancy test was performed when necessary to exclude pregnancy.

Exclusion Criteria:

* Patients with type 1 diabetes, gestational diabetes or other special type of diabetes;
* All kinds of acute complications such as diabetic ketoacidosis and non-ketohyperosmotic syndrome were screened in the first month;
* Patients who had received other stem cell therapy before screening;
* Patients with poorly controlled hypertension had a blood pressure of 160/100mmHg during screening;
* Screening those who had taken thiazolidinedione, DDP-IV inhibitors and GLP-1 drugs within the first 3 months;
* Insulin therapy was used for less than 1 year before screening, and only subcutaneous injection was performed daily for nearly 3 months; One dose insulin;
* Patients with pancreatic diseases, including those with acute and chronic pancreatitis and pancreatic tumors;
* Those with other malignant or suspected tumor tendencies;Or in active phase of infection (including hepatitis b or HCV);Immunodeficiency virus (HIV) positive patients;
* Patients suffering from other serious systemic diseases (such as cardiovascular system, respiratory system, digestive system, nervous system, endocrine system, genitourinary system, immune system and blood system);
* Patients with abnormal liver and kidney function, such as serum bilirubin TBIL exceeding 1.5 times of the normal upper limit, glutamate AST and ALT exceeding 2.5 times of the normal upper limit, and serum creatinine Cr exceeding 1.2 times of the normal upper limit;
* Being treated with systemic sex hormones (glucocorticoids), immunosuppressive or cytotoxic agents;
* Disabled person (blind, deaf, dumb, mentally handicapped, or physically disabled) as prescribed by law, a pregnant and lactating woman;People with mental illness;Patients who have a history of drug abuse or alcohol dependence within 5 years;
* Patients with contraindications or allergies treated in this study;
* Subjects who participated in other clinical studies within the last three months.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Total daily insulin | 1 week
  After treatment total daily insulin dose changes

SECONDARY OUTCOMES:
HbAlc | 1 week
  The proportion of patients with HbA1c < 7.0% and < 6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Qin Huang, Doctor, Principal Investigator — Changhai houspital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No